CLINICAL TRIAL: NCT00196469
Title: Randomized Double Blind Trial Comparing Heparin and Placebo as Additives to Continuous Infusion in Intensive Care Neonates for Prevention of Ventilation
Brief Title: Impact of Heparin on the Need for Mechanical Ventilation in Neonates
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EMAU16253.00.00
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2006-09

CONDITIONS: Respiration, Artificial; Hemorrhage
MeSH Terms: conditions — Respiratory Aspiration; Hemorrhage | interventions — Heparin

INTERVENTIONS:
Drug: heparin

SUMMARY:
This study is designed to test an incidental finding of a previous trial in which post hoc analysis showed that the rate of intensive care newborns requiring mechanical ventilation was lower in the group receiving heparin with the continuous infusion as compared to the placebo group.

DETAILED DESCRIPTION:
Title: Randomized double blind trial comparing heparin and placebo as additives to continuous infusion in intensive care neonates for prevention of mechanical ventilation

Primary endpoint: Percentage of neonates requiring mechanical ventilation in both groups

Secondary endpoints: Duration of dependency on mechanical ventilation; major bleedings, incidence of heparin-induced thrombocytopenia and of anti-platelet factor 4/heparin antibodies

ELIGIBILITY:
Inclusion Criteria:

* Newborns < day 28 of life
* Necessity for intensive care treatment
* Necessity for parenteral drug or fluid application for at least five days
* Informed consent of parents

Exclusion Criteria:

* Body weight < 500g
* Mechanical ventilation directly after birth
* Major malformations
* Absolute indication for heparin
* Inborn hemorrhagic disease (e.g. hemophilia, von Willebrand disease)
* Cerebral bleeding or other major bleeding
* Platelet count < 50,000/µl

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2003-12; Study Completion 2007-03

PRIMARY OUTCOMES:
percentage of neonates requiring mechanical ventilation

SECONDARY OUTCOMES:
duration of dependency on mechanical ventilation
major bleeding
heparin induced thrombocytopenia
anti PF4/heparin antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Greinacher, MD, Study Chair — Institute for Immunology and Transfusion Medicine, Ernst-Moritz-Arndt-University Greifswald; Christoph Fusch, MD, Study Director — Pediatric Department, Ernst-Moritz-Arndt-University Greifswald; Anne F Klenner, MD, Principal Investigator — Medical Faculty, Ernst-Moritz-Arndt University Greifswald
Locations (1):
- University Hospital Department of Pediatrics/Institute for Immunology and Transfusion Medicine, Greifswald, Germany